CLINICAL TRIAL: NCT01914718
Title: Dose-adjusted EPOCH-R in Patients With Diffuse Large B-cell Lymphoma: a Phase II Study
Brief Title: Dose-adjusted EPOCH-R in MYC Positive DLBCL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual of eligible patients
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ye Guo, Dr., Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMTG 13-02
Record Dates: First submitted 2013-03-02; First posted 2013-08-02 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: DLBCL; DA-EPOCH-R
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DA-EPOCH-R (Experimental): rituximab 375mg/m2 IV day 0, etoposide 50mg/m2/d CIV days 1-4, doxorubicin 10mg/m2/d CIV days 1-4, vincristine 0.4mg/m2/d CIV days 1-4, cyclophosphamide 750mg/m2 IV day 5, prednisone 50mg PO days 1-5 twice per day
  Interventions: Drug: DA-EPOCH-R

INTERVENTIONS:
Drug: DA-EPOCH-R — rituximab 375mg/m2 IV day 0, etoposide 50mg/m2/d CIV days 1-4, doxorubicin 10mg/m2/d CIV days 1-4, vincristine 0.4mg/m2/d CIV days 1-4, cyclophosphamide 750mg/m2 IV day 5, prednisone 50mg PO days 1-5 twice per day
  Other Names: mabthera

SUMMARY:
The aim of this study is to evaluate the efficacy and toxicity of dose-adjusted EPOCH-R in patients with MYC positive diffuse large B-cell lymphoma.

DETAILED DESCRIPTION:
The prognosis of MYC positive diffuse large B-cell lymphoma (DLBCL) is very poor even treated with R-CHOP regimen. Recently, dose-adjusted EPOCH-R was shown to be effective in patients with DLBCL and relapsed/refractory Burkitt lymphoma. The aim of this study is to evaluate the efficacy and toxicity of dose-adjusted EPOCH-R in patients with MYC positive diffuse large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated MYC positive diffuse large B-cell lymphoma
* Age range 18-70 years old
* Eastern Cooperative Oncology Group performance status 0-2
* Life expectancy of more than 3 months
* Adequate organ function

Exclusion Criteria:

* Primary or secondary central nervous system involvement
* Previous serious cardiac disease
* History of other malignancies except cured basal cell carcinoma of skin and carcinoma in-situ of uterine cervix
* Pregnant or lactating women
* Serious uncontrolled diseases and intercurrent infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
3-year progression-free survival | 3 years

SECONDARY OUTCOMES:
Objective response rate | 4 months
3-year overall survival | 3 years
Toxicity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China